CLINICAL TRIAL: NCT04019015
Title: A Prospective Randomized Prehospital Trial Comparing Kcentra Plus Standard of Care to Standard of Care Alone in Trauma Patient With Hemorrhagic Shock
Brief Title: Prehospital Kcentra for Hemorrhagic Shock
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Martin A Schreiber, MD, Professor and Chief of Trauma, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OHSU IRB 17077
Record Dates: First submitted 2019-06-02; First posted 2019-07-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Trauma Injury
Keywords: Shock, Hemorrhagic; Trauma; Mortality; Wounds and Injuries; Hemorrhage
MeSH Terms: conditions — Accidental Injuries; Shock, Hemorrhagic; Wounds and Injuries; Hemorrhage | interventions — Factor IX

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Kcentra (Experimental): A single dose of Kcentra based on estimated body weight
  * 2000 U for patients with an estimated body weight ≤ 75kg
  * 3000 U for patients with an estimated body weight > 75kg
  Interventions: Drug: Prothrombin Complex Concentrate, Human
- Placebo (Placebo Comparator): A single infusion of volume matched placebo solution (Normal Saline)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prothrombin Complex Concentrate, Human — Prothrombin Complex Concentrate (PCC) prepared from human plasma and contains blood coagulation factors
  Other Names: Kcentra
  Arms: Kcentra
Drug: Placebo — Normal saline solution
  Arms: Placebo

SUMMARY:
This is a pilot trial being performed to evaluate the feasibility, to include the ability of EMS to identify patients in shock and the ability to package, store, and administer Kcentra in the field.

DETAILED DESCRIPTION:
Prospective randomized trials have shown that 4-factor prothrombin complex concentrate (4FPCCs) result in more rapid correction of coagulopathy and greater likelihood of achieving hemostasis in patients receiving vitamin K antagonists who require emergent operations or who are bleeding. 4FPCCs have not been studied in the pre-hospital setting as a primary resuscitative adjunct. The investigators believe the effects of Kcentra to prevent or treat coagulopathy early after injury combined with its ability to treat the endotheliopathy of trauma and prevent organ failure will results in improved outcomes in severely injured trauma patients with hemorrhagic shock. The investigators have chosen to study a population of trauma patients in severe hemorrhagic shock (SBP < 70mmHg) because this population is at greatest risk for developing acute coagulopathy of trauma and has the greatest potential to benefit from the proposed therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Trauma patients age 18 years or greater, or weight > 50 kg if age unknown
2. Systolic blood pressure < 70 mmHg
3. Suspicion of hemorrhagic shock based on mechanism of injury
4. EMS transport to a participating trauma center

Exclusion Criteria:

1. Age less than 18
2. Unknown time of injury
3. Out-of-hospital cardiopulmonary resuscitation
4. Known history of thromboembolic disorders or stroke or suspicion by EMS of a recent stroke
5. Known oral anti-coagulant use to include warfarin and novel anti-coagulants
6. Severe hypothermia (<28°C)
7. Drowning or asphyxia due to hanging
8. Burns more than 20% total body surface area
9. Evidence of devastating blunt traumatic brain injury to include fixed and dilated pupils, asymmetric pupils and extrusion of brain matter
10. Isolated blunt or penetrating head injury
11. Isolated spinal cord injury
12. Ground level (same level) falls
13. Inability to obtain intravenous access
14. Inability to administer randomized therapy within 4 hours of ambulance notification
15. Known transfers and inter-facility transfers
16. Known Do Not Resuscitate (DNR) prior to randomization
17. Known or suspected pregnancy
18. Known prisoners
19. Patients who have activated the "opt-out" process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of study drug administration | First 24 hours after injury
  Number of study drug kits opened and given to patients prior to hospital arrival.

SECONDARY OUTCOMES:
Mortality | First 30 days after injury
  To evaluate mortality at 3 hour, 24 hour, and 30 days
Hospital Free Days | First 30 days after injury
  Number of days out of the hospital
ICU Free Days | First 30 days after injury
  Number of days out of the ICU
Ventilator Free Days | First 30 days after injury
  Number of days not on a ventilator
Blood Transfusions | First 24 hours after injury
  The amount of blood products transfused in the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Schreiber, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No